CLINICAL TRIAL: NCT01585623
Title: An Open-label, Two-treatment Crossover Pharmacokinetic Interaction Study of Repeated Doses of SAR302503 on Pharmacokinetics of a Single Dose Cocktail of Omeprazole, Metoprolol, and Midazolam Used as Probe Substrates for CYP2C19, CYP2D6 and CYP3A4 Activities, Respectively in Adult Patients With Refractory Solid Tumors
Brief Title: Drug Interaction Study of SAR302503 in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INT12497; U1111-1125-8930 (Other: UTN)
Record Dates: First submitted 2012-04-13; First posted 2012-04-26 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2013-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — fedratinib; Omeprazole; Metoprolol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Segment 1 (Experimental): two single doses of omeprazol/metoprolol/midazolam on day-1 and day 15 without food, SAR302503 500 mg once daily without food for 15 days
  Interventions: Drug: SAR302503; Drug: omeprazol; Drug: metoprolol; Drug: midazolam
- Segment 2 (Experimental): SAR302503 500 mg once daily without food in 28-day per cycle
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral
Drug: omeprazol — Pharmaceutical form:capsule
  Route of administration: oral
  Arms: Segment 1
Drug: metoprolol — Pharmaceutical form:tablet
  Route of administration: oral
  Arms: Segment 1
Drug: midazolam — Pharmaceutical form:solution
  Route of administration: oral
  Arms: Segment 1

SUMMARY:
Primary Objective:

* To assess the effect of 15-day repeated oral doses of 500 mg SAR302503 on the cytochrome P450 activity using a CYP probe cocktail (2C19, 2D6 and 3A4).
* To document pharmacokinetics of SAR302503 after repeated 500 mg oral daily doses.

Secondary Objectives:

* To assess the safety profile of 15-day repeated oral doses of 500 mg SAR302503 in Segment 1
* To characterize the safety and tolerability of 28-day consecutive doses of 500 mg SAR302503 in Segment 2
* To determine antitumor activity in Segment 2

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a period to assess eligibility (screening period 21 days), followed by a treatment period of at least 15 days of study treatment, and an end-of-treatment visit at least 30 days following the last administration of study drug. However, treatment may continue if patients are receiving benefit and do not have unacceptable toxicity or meet study withdrawal criteria.

ELIGIBILITY:
Inclusion criteria :

* Histologically or cytologically confirmed advanced solid malignancy that is metastatic or unresectable, and for which standard curative measures do not exist
* Signed informed consent

Exclusion criteria:

* Less than 18 years of age.
* Limited physical functioning (as evaluated by the Eastern Cooperative Oncology Group (ECOG) scale)
* Inability to follow study requirements and schedule
* Treatment of cancer within 3 weeks of study, concurrent treatment in another clinical trial or with any other anti-cancer therapy
* Serious medical illness at same time of study and/or significantly abnormal lab reports
* Lack of pregnancy contraception (women of childbearing potential), pregnancy, or breast feeding.
* Men who partner with a woman of childbearing potential, unless they agree to use effective contraception while on study drug
* Continued toxic effects of prior chemotherapy
* Evidence of other concurrent active malignancy
* Other concurrent serious illness or medical condition
* Cardiac abnormalities include bradycardia, AV block or other conduction defect on ECG, and patients taking a beta blocker.
* Patients with Insulin-Dependent Diabetes Mellitus.
* Patients with known active (acute or chronic) hepatitis A, B, C, and hepatitis B and C carries. Prior history of chronic liver disease (e.g., chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH]).
* Inadequate organ function
* History of partial or total gastrectomy, or, if in the opinion of the investigator, have any other disorder that would inhibit absorption of oral medications.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Omerprazole/metoprolol/midazolam - Pharmacokinetic parameter: AUC, AUClast | predose and up to 24 hours post dose on Days -1, 1, 15 and 16

SECONDARY OUTCOMES:
Omerprazole/metoprolol/midazolam - Pharmacokinetic parameter : Cmax, Tmax, and t1/2z | predose and up to 24 hours post dose on Days -1, 1, 15 and 16
SAR302503 - Pharmacokinetic parameter : Cmax, Tmax, Ctrough and AUC0-24 | Day-1 to Day 16
Clinical and laboratory events graded by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v4.03 (Segment 1 and 2) | up to maximum 2 years
Objective response ratio (Complete response (CR) and partial response (PR)) (Segment 2) | up to 2 cycles ( i.e. 10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840004, Augusta, Georgia
  - Investigational Site Number 840001, Detroit, Michigan
  - Investigational Site Number 840002, Philadelphia, Pennsylvania